CLINICAL TRIAL: NCT06250595
Title: European Rare Blood Disorders Platform (ENROL)
Acronym: ENROL
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: ERN-EuroBloodNet (European Reference Network on Rare Hematological Diseases (Unknown)
Responsible Party: Sponsor
Other Study IDs: PR(AMI)294/2022
Record Dates: First submitted 2023-12-04; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-12

CONDITIONS: Anemia; Bone Marrow Failure; Bleeding Disorder; Iron Metabolism Disorders; Myeloma; Lymphoid Neoplasm; Myeloma, Malignant; Leukemia; Anemia, Sickle Cell; Thalassemia; Blood Cancer; Red Cell Membrane and Enzyme Abnormalities
Keywords: Anemia; Bone Marrow Failure; Bleeding disorder; Iron metabolism disorder; Myeloid; Lymphoid; Blood cancer; Leukemia; Red Cell membrane and Enzyme Abnormalities; Thalassemia; Sickle Cell Disease
MeSH Terms: conditions — Anemia; Bone Marrow Failure Disorders; Hemostatic Disorders; Iron Metabolism Disorders; Neoplasms, Plasma Cell; Leukemia; Anemia, Sickle Cell; Thalassemia; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Inherited Rare Anaemia Disorders, including inherited Bone Marrow Failures: Patients with Inherited Rare Anemia Disorders, including inherited Bone Marrow Failures, stratified by gender, age, and/or variants/types if applicable.
  Interventions: Other: Collection of clinical and laboratory data from EHR.
- Acquired Bone Marrow Failures: Patients with Acquired Bone Marrow Failures, stratified by gender, age, and/or variants/types if applicable.
  Interventions: Other: Collection of clinical and laboratory data from EHR.
- Rare bleeding-coagulation disorders and related diseases: Patients with Rare bleeding-coagulation disorders and related diseases, stratified by gender, age, and/or variants/types if applicable.
  Interventions: Other: Collection of clinical and laboratory data from EHR.
- Hemochromatosis and other rare genetic disorders of iron metabolism and heme synthesis: Patients with hemochromatosis and other rare genetic disorders of iron metabolism and heme synthesis, stratified by gender, age, and/or variants/types if applicable.
  Interventions: Other: Collection of clinical and laboratory data from EHR.
- Myeloid malignancies: Patients with Myeloid malignancies, stratified by gender, age, and/or variants/types if applicable.
  Interventions: Other: Collection of clinical and laboratory data from EHR.
- Lymphoid malignancies: Patients with lymphoid malignancies, stratified by gender, age, and/or variants/types if applicable.
  Interventions: Other: Collection of clinical and laboratory data from EHR.

INTERVENTIONS:
Other: Collection of clinical and laboratory data from EHR. — Observational sutdy

SUMMARY:
ENROL, the European Rare Blood Disorders Platform has been conceived in the core of ERN-EuroBloodNet as an umbrella for both new and already existing registries on Rare Hematological Diseases (RHDs). ENROL aims at avoiding fragmentation of data by promoting the standards for patient registries' interoperability released by the EU RD platform.

ENROL's principle is to maximize public benefit from data on RHDs opened up through the platform with the only restriction needed to guarantee patient rights and confidentiality, in agreement with EU regulations for cross-border sharing of personal data.

Accordingly, ENROL will map the EU-level demographics, survival rates, diagnosis methods, genetic information, main clinical manifestations, and treatments in order to obtain epidemiological figures and identify trial cohorts for basic and clinical research. To this aim, ENROL will connect and facilitate the upgrading of existing RHD registries, while promoting the building of new ones when / where lacking. Target-driven actions will be carried out in collaboration with EURORDIS for educating patients and families about the benefits of enrolment in such registries, including different cultural and linguistic strategies.

The standardized collection and monitoring of disease-specific healthcare outcomes through the ENROL user-friendly platform will determine how specialized care is delivered, where are the gaps in diagnosis, care, or treatment and where best to allocate financial, technical, or human resources.

Moreover, it will allow for promoting research, especially for those issues that remain unanswered or sub-optimally addressed by the scientific community; furthermore, it will allow promoting clinical trials for new drugs. ENROL will enable the generation of evidence for better healthcare for RHD patients in the EU as the ultimate goal.

ENROL officially started on 1st June 2020 with a duration of 36 months. ENROL is co-funded by the Health Programme of the European Union under the call for proposals HP-PJ-2019 on Rare disease registries for the European Reference Networks. GA number 947670

DETAILED DESCRIPTION:
Study Title:

European Rare Blood Disorders Platform (ENROL)

Study Objectives:

The European Rare Blood Disorders Platform (ENROL) is conceived in the core of the European Reference Network on Rare Hematological Diseases (ERN-EuroBloodNet), as the umbrella platform for both new and already existing registries on Rare Hematological Diseases (RHDs) avoiding fragmentation of data by promoting the interoperability standards for patient registries.

ENROL aims at mapping demographics, diagnosis methods, genetic data, main clinical manifestations and treatments at the EU level by enabling the connection, upgrading and building of EU patients registries in line with EU data protection and interoperability standards with the following major objectives:

Promoting research: allowing the identification of patient cohorts to facilitate the development of collaborative projects on basic and clinical research on RHD Epidemiological surveillance: pooling of available data on registries and databases across European countries to monitor trends and provide essential epidemiologic information on RHD while enabling the generation of evidence for the optimum allocation of resources and health planning For this, ENROL will obtain comparable EU data for RHD on demographics, survival rates, diagnosis methods, genetic information, main clinical manifestations and treatments by promoting the interoperability standards for patient registries in line with the European Platform on Rare Disease Registration (EU RD Platform). ENROL is officially endorsed by the European Hematology Association (EHA).

Methodology:

Data on patients with RHDs will be collected retrospectively and prospectively at the time of inclusion on the registry and at 12-month intervals for all registered patients.

The ENROL strategy for data gathering combines the exhaustiveness of data collection at EU level for health planning and epidemiological purposes, with a higher level of RHD data granularity for promoting research and identification of patients' cohorts.

Accordingly, the platform has been designed to integrate data from any available sources, including Healthcare providers (ERN-EuroBloodNet members / Other EU healthcare providers) and EU/national/local existing registries. Data entry is also allowed with different levels of granularity to pursue ENROL aims, including counts/aggregated level data to increase data exhaustiveness at the EU level required for the epidemiological surveillance, and pseudonymised individual level data to promote research and facilitate the identification of trial groups.

As defined in GDPR Art. 26, a Joint Controllership is being established where the institutions conforming the Consortium (HUVH/VHIR, ULB/ERASME, CING and AP-HP) for the jointly determine the purposes and means of processing and assume equal responsibilities in terms of data protection.

Data processing and analyses will be conducted in various sub studies, after every 1000 patients included in the European Registry and/or at the end of each interim follow-up period (every 12 months).

Disease coverage

The study population consist of both males and females aged from 0 to 100 year old diagnosed as RHD according to ORPHANET classification (ORPHA 97992), including myeloid and lymphoid tumors (ORPHA 68347), rare anaemia disorders (ORPHA 108997), rare coagulation disorders (ORPHA 98429), and polycythemia (ORPHA 98427), and further complemented with rare hereditary hemochromatosis (ORPHA220489), included in the disease scope of ERN-EuroBloodNet following a request from well-established patient groups and experts.

Accordingly, ENROL disease coverage results in more than 450 different entities with differential clinical and etiological features i.e. oncological vs non-oncological, hereditary vs acquired, or significant difference frequency, among others, which can be classified into the following disease groups:

RAD: Inherited Rare Anaemia Disorders, including inherited Bone Marrow Failures BMF: Acquired Bone Marrow Failures Bleeding: Rare bleeding-coagulation disorders and related diseases HH-Iron: Hemochromatosis and other rare genetic disorders of iron metabolism and heme synthesis Myeloid: Myeloid malignancies Lymphoid: Lymphoid malignancies

ENROL dataset has been conceived in a bottom-up design for ensuring the capture of the common elements for rare diseases in line with the EU recommendations and with the EU RD platform, and the key features common for the whole spectrum for RHDs. Furthermore, the latest level can be stepped up for the definition of domain specific elements that support the in-depth analysis.

In the spirit of ENROL aims to promote the connection and linkage of available data sources and the creation of new registries where lacking. ENROL promotes collaborations for supporting the a) upgrade the existing registries and b) create new European registries in compliance with the standards of interoperability and ENROL policy. Collaboration agreements will be in place for the transfer of a subset of the data elements gathered to ENROL.

Study Duration and funding

An extensive recruitment period and follow-up, as well as geographical coverage, is desirable for long-term sustainability of the European Epidemiological Platform. Accordingly, ENROL has not an expected ending date but continue the pooling and processing of data for an indeterminate period of time.

ENROL is co-funded by the Health Programme of the European Union under the call for proposals HP-PJ-2019 on Rare disease registries for the European Reference Networks. GA number 947670.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to be included in the ENROL Registry
* Age from 0-100, both female and male
* Diagnosed as RHDs according to ORPHANET classification
* Able and willing to provide written informed consent (patient or legal representative for minors) if needed according to national legislation.

Exclusion Criteria:

* Patients diagnosed as traits or trait conditions for other recessive RHDs

Max Age: 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Rare Hematological Disease
Sampling Method: Probability Sample
Enrollment: 37090 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2037-07 (Estimated); Study Completion 2037-07 (Estimated)

PRIMARY OUTCOMES:
Demography and epidemiology | 15 years
  To collect and to describe demographics and epidemiological data of any type of RHDs.

CONTACTS AND LOCATIONS:
Overall Officials: María del Mar Manú Pereira, PhD, Principal Investigator — Vall d'Hebron Institut de Recerca / University Hospital Vall d'Hebron (VHIR / HUVH); Béatrice Gulbis, MD, Principal Investigator — Hôpital ERASME / ULB (ERASME_ULB); Petros Kountouris, PhD, Principal Investigator — Cyprus Institute of Neurology and Genetics (CING); Pierre Fenaux, MD, Principal Investigator — Assistance Publique - Hopitaux de Paris (AP-HP)
Locations (1):
- María del Mar, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: EU EurobloodNet offficial Website — https://eurobloodnet.eu/
- See also: European Commission website section on European Reference Networks — https://health.ec.europa.eu/european-reference-networks/overview_en
- See also: EU ENROL Official Website — https://eurobloodnet.eu/enrol-first/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT06250595/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT06250595/ICF_001.pdf